CLINICAL TRIAL: NCT06374264
Title: A Single Arm, Prospective, Multi-Center, Feasibility Study to Evaluate the Acceptability and Safety of MR-C-014 in Persons With Neuromyelitis Optica Spectrum Disorder (NMOSD) Who Have an Impaired Gait
Brief Title: Acceptability and Safety of MR-C-014 in Persons With Neuromyelitis Optica Spectrum Disorder
Acronym: aNiMatO
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: MedRhythms, Inc. (Industry)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NM100
Record Dates: First submitted 2024-04-10; First posted 2024-04-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: Rhythmic Auditory Stimulation (RAS); Neurology
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention (Experimental): Participants will be asked to use MR-C-014 for 24 sessions (30 minutes each), 3 times a week for 8 weeks.
  Interventions: Device: MR-C-014

INTERVENTIONS:
Device: MR-C-014 — Use of device 3 times per week (for 30 minutes) for 8 weeks - for a total of 24 sessions.

SUMMARY:
The purpose of this proof of concept study is to assess the acceptability and safety of MR-C-014 in persons with Neuromyelitis optica spectrum disorder (NMOSD) who have a gait deficit.

DETAILED DESCRIPTION:
This is a single arm, prospective, multi-center feasibility study designed to evaluate the acceptability and safety of MR-C-014.

MR-C-014 is an autonomous neurorehabilitation system based on the principles of Rhythmic Auditory Stimulation (RAS) and is designed to operate digitally and autonomously. The core mechanism of RAS is "auditory-motor entrainment." Studies have shown that there is rich connectivity between the auditory and motor systems via multiple cortical and subcortical networks.

The MR-C-014 system consists of two foot sensors that measure walking, a locked touchscreen device preloaded with a proprietary software application, a headset, and charging equipment. The electronic components are powered by lithium-ion rechargeable batteries.

MR-C-014 is an investigational device.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years of age (inclusive).
2. Able to read and/or understand English.
3. Meets revised diagnostic criteria for NMOSD proposed by the International Panel for NMO Diagnosis (IPND) in 2015.
4. Past clinical history of Transverse Myelitis as seen on imaging or as determined by clinical review by the investigator.
5. Demonstrates an observable gait deficit resulting from a diagnosis of NMOSD as determined by the Investigator or medical history review.
6. Currently able to walk at a speed greater or equal to 0.4 m/s, but less than 1.5 m/s, as determined by walking speed during a Timed 25-Foot Walk Test (T25FWT) (cane(s), walking stick(s), crutch(es), wheeled walker, external functional neuromuscular stimulator(s), and ankle foot orthosis allowed).

   a. Note: if assistive devices are planned to be used during the Intervention Phase walking sessions, they should be used during the Screening, Baseline, and Closing visit gait assessments as well.
7. Has a reciprocal gait pattern.

   a. Note: a non-reciprocal gait pattern is defined as a 3-point step pattern. Participants must have a 2-point step pattern to qualify. Asymmetry seen in gait is acceptable.
8. Ability and willingness to provide Informed Consent.

Exclusion Criteria:

1. Unable or unwilling to comply with study protocol.
2. People who become pregnant or are pregnant (due to expected changes in gait patterns).
3. Unable to safely participate in protocol-defined walking sessions of 30-minute duration as determined by the investigator.
4. Significant co-morbid medical or neurological disease or injury, or treatment for such conditions that currently affects, or has potential to affect, participant gait for safety during participation in the study as determined by the investigator.
5. Has an external lower limb prosthetic ("artificial limb").
6. Initiated physical therapy for lower limb in the past 4 weeks or anticipated to start due to safety concerns (e.g., falls).
7. Requires at least one seated rest during the T25FWT.
8. Initiation, change, or discontinuation of disease-modifying therapy in the past 3 months known to affect gait (e.g., dalfampridine, corticosteroid, medications for spasticity).
9. Recent NMOSD relapse (last 3 months) and/or hospitalization.
10. Severe hearing impairment with or without the use of hearing aids, such that the participant cannot hear the rhythmic music stimulus consistently, as determined by participant and investigator.
11. Treatment with a gait-based investigational intervention within the last 3 months. Enrollment in observational studies is allowed.
12. Vulnerable populations as deemed inappropriate for study by investigator. For this protocol, vulnerable persons are considered to be those who are relatively (or absolutely) incapable of protecting their own interests.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Participant acceptability of MR-C-014 | Intervention period (of up to 8 weeks)
  Assesses participant engagement via logged use of MR-C-014
Number of device-related adverse events (AEs) | Weekly for up to 8 weeks
  Assesses the safety of MR-C-014 in NMOSD patients with a gait deficit

SECONDARY OUTCOMES:
6-Minute Walk Test (6MWT) | Baseline and closing (up to 8 weeks)
  Assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance (distance in meters)
Number of walks per week | Weekly for up to 8 weeks
  Assesses adherence to recommended frequency of MR-C-014 use. Recommended frequency is 3 walks per week for 8 weeks.

OTHER OUTCOMES:
Spatiotemporal symmetry of gait as measured by the MR-C-014 sensors | Baseline and closing (up to 8 weeks)
  Assesses spatiotemporal symmetry of gait in NMOSD patients with a gait deficit while using MR-C-014
Spatiotemporal variability of gait as measured by the MR-C-014 sensors | Baseline and closing (up to 8 weeks)
  Assesses spatiotemporal variability of gait in NMOSD patients with a gait deficit while using MR-C-014
Stride length as measured by the MR-C-014 sensors | Baseline and closing (up to 8 weeks)
  Assesses stride length in NMOSD patients with a gait deficit while using MR-C-014
Falls Efficacy Scale-International (FES-I) | Baseline and closing (up to 8 weeks)
  A 16-item self-administered questionnaire designed to assess fear of falling in mainly community-dwelling older population. Minimum score = 16 (no concern about falling); maximum score = 64 (severe concern about falling).
Number of falls as recorded in Falls Diary | Weekly for up to 8 weeks
  Assesses number of falls in NMOSD patients with a gait deficit
Multiple Sclerosis Walking Scale (MSWS-12) | Baseline and closing (up to 8 weeks)
  A self-report measure of the impact of MS on the individual's walking ability. Minimum score = 12 (not at all impacted); maximum score = 60 (extremely impacted).
Visual Analogue Scale (VAS) | Baseline and closing (up to 8 weeks)
  A validated, subjective measure to assess pain intensity. Minimum score = 0 (no pain); maximum score = 10 (worst pain possible).
Generalized Anxiety Disorder-7 (GAD-7) | Baseline and closing (up to 8 weeks)
  A self-administered patient questionnaire used as a screening tool and severity measure for generalized anxiety disorder. Minimum score = 0 (no anxiety); maximum score = 21 (severe anxiety).
9 Hole Peg Test (9-HPT) | Baseline and closing (up to 8 weeks)
  A standardized, quantitative assessment used to measure finger dexterity (time in seconds).
Symbol Digit Modalities Test (SDMT) | Baseline and closing (up to 8 weeks)
  A measure of cognitive processing speed. Minimum score = 0; maximum score = 110. Higher score indicates faster processing speed.
Fatigue Scale for Motor and Cognitive Functions (FSMC) | Baseline and closing (up to 8 weeks)
  A 20-item scale developed as a measure of cognitive and motor fatigue for people with MS. Minimum score = 20; maximum score = 100. Higher score indicates higher level of fatigue.
Expanded Disability Status Scale (EDSS) Ambulation Score | Baseline and closing (up to 8 weeks)
  The EDSS is a scale for assessing the level of disability in people with multiple sclerosis The ambulation score specifically assesses impairment to ambulation. Minimum score = 0; maximum score = 10. Higher score indicates greater disability.
Activities-Specific Balance Confidence Scale (ABC) | Baseline and closing (up to 8 weeks)
  A self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness. Minimum score = 0 (no confidence); maximum score = 100 (complete confidence).
Patient Experience and Satisfaction Survey | Closing (at up to 8 weeks)
  Assesses patient satisfaction with the MR-C-014 device

CONTACTS AND LOCATIONS:
Overall Officials: Eric Klawiter, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Sheperd Center, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No